CLINICAL TRIAL: NCT03389100
Title: Tau Positron Emission Tomography (PET) Imaging in the Northern Manhattan Study of Metabolism and Mind (NOMEM) With 18F-MK6240.
Brief Title: Tau PET Imaging in the Northern Manhattan Study of Metabolism and Mind.
Acronym: NOMEM-Tau
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Hebrew Home at Riverdale (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, José A. Luchsinger, Associate Professor, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAR1419b; R01AG050440 (NIH); R01AG055299 (NIH); RF1AG051556 (NIH)
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2; Pre-diabetes
Keywords: diabetes; hyperglycemia; tau
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Diabetes Mellitus; Hyperglycemia; Pick Disease of the Brain | interventions — MK-6240

STUDY DESIGN:
Intervention Model Description: Study subjects will receive a single injection of 18F-MK6240 for tau positron emission tomography (PET) imaging two times, separated by an interval between 18 and 30 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-MK6240 injection (Experimental): intravenous injection of 18F-MK-6240, up to 5 mCi (185 MBq), IV, total of one injection per PET scan (2 injections in total with an interval of 18 to 30 months)
  Interventions: Drug: 18F-MK6240 injection

INTERVENTIONS:
Drug: 18F-MK6240 injection — Intravenous injection of 18F-MK-6240, up to 5 mCi (185 MBq), total of one injection per PET scan (2 injections in total with an interval of 18 to 30 months)
  Other Names: MK6240

SUMMARY:
This is a single center brain Positron Emission Tomography (PET) study of 18F-MK-6240. Eligible participants are persons from Northern Manhattan who self-identify as Hispanic, non-Hispanic Black, or Non-Hispanic White, who are 55 to 69 years of age, of both sexes, without dementia, who have already agreed to undergo, of have undergone, brain amyloid PET and magnetic resonance imaging (MRI). Those eligible will have one brain PET scan with 18F-MK-6240, repeated after 18 months to 30 months. Vital signs will be checked prior to injection of 18F-MK-6240 and again at the completion of the PET scan. The primary objective is to relate diabetes status and glycemia to in-vivo brain tau accumulation, across and within ethnic and racial groups.

DETAILED DESCRIPTION:
1. Subject recruitment and screening procedures. Subjects will be recruited from community dwelling persons from Northern Manhattan, men and women, aged 55 to 69 years, who have already undergone or agreed to undergo, brain magnetic resonance imaging (MRI) and Florbetaben positron emission tomography (PET) as part of Columbia IRB protocol AAAQ2950 (PI: Luchsinger). Recruitment of participants for these studies and all study procedures, including brain MRI, Florbetaben PET, and tau PET, are funded by existing grant from the National Institutes of Health awarded to PI Luchsinger (R01AG050440, RF1AG051556-01S2, R01AG055299)
2. Imaging procedures related to 18F-MK-6240 PET. One brain MRI will be performed on each subject using a 3 T Philips scanner. Sequences performed will include 3D T1 (MPRAGE, 180 slice 1 mm resolution, 256 x 256 voxel count) for volumetric analysis and clinical sequences to exclude subjects with significant intracranial pathology unrelated to AD, such as malignant brain tumor of subdural hematoma. PET scans will take place on a Biograph mCT PET scanner (Siemens Healthcare) at the CUMC Kreitchman PET Center. Subjects will have one PET scan with 18F-MK-6240 (injected activity up to 5 mCi = 185 MBq). PET imaging will be performed without arterial sampling. Vital signs (blood pressure, heart rate, respiratory rate, and temperature) will be checked prior to injection of 18F-MK-6240, then at the completion of the PET scan. 18F-MK-6240 will be purchased from Cerveau Technologies, Inc. via a licensed production facility. Subjects will not be informed of 18F-MK-6240 PET scan results, as this scan is used only in research and have not yet been validated for clinical use. Subjects will be informed if a clinically important abnormality is detected on MRI or PET imaging (e.g., brain tumor).
3. Image processing FreeSurfer (http://surfer.nmr.mgh.harvard.edu/), the MRI software package comprising a suite of automated tools for segmentation, reconstruction, and derivation of regional volumes and surface-based rendering, will be used for derivation of regions-of-interest (ROIs). Eleven ROIs will be extracted from the structural T1 image: entorhinal cortex, hippocampus, inferior temporal cortex, combined superior and middle temporal cortex, superior parietal lobule, inferior parietal lobule, precuneus, occipital cortex, prefrontal cortex, striatum, and thalamus. 18F-MK-6240 PET images will be analyzed as follows: Freesurfer based ROIs will be applied to coregistered PET images. Correction for partial volume effects using a region-based voxel-wise method92 will be applied to compare to partial volume uncorrected data. Regional time-activity curves will be extracted from the PET scans, including cerebellum which will be used as a reference region. Standardized uptake value ratio (SUVR) values will be calculated by dividing SUV values for each target region by that of the cerebellum. Alternative analytic methods such as Logan DVR and Simplified Reference Tissue Method may also be applied to compare to SUVR data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 to 69 years
2. Without dementia
3. Fluent in English and/or Spanish.
4. Living in Northern Manhattan.
5. Self-identified as Hispanic, non-Hispanic Black, or non-Hispanic White.
6. Already had or agreed to have a brain MRI and Florbetaben PET.
7. Able to participate in all scheduled evaluations and to complete all required tests and procedures.

Exclusion Criteria:

1. Dementia diagnosis
2. Certain significant medical conditions, which make study procedures of the current study unsafe. Such serious medical conditions include uncontrolled epilepsy and multiple serious injuries.
3. Persons with serious chronic conditions (e.g. Liver Cirrhosis, renal failure), which, in the opinion of the investigator, could increase the risk of un-anticipated adverse events.
4. Contraindication to MRI scanning
5. Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
6. Inability to have a catheter in subject's vein for the injection of radioligand.
7. Inability to have blood drawn from subject's veins.
8. Women in the age group that we are recruiting are highly unlikely to be pre-menopausal, and thus, highly unlikely to be menstruating. However, we will ask all women if they are post-menopausal, and in the rare case that they are not, we will conduct a urine pregnancy test to rule out pregnancy.

Breastfeeding women will be excluded, although we expect this situation to be rare

Ages: 55 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
18F-MK6240 standardized update value ratio (SUVR) | 18 to 30 months
  The primary outcome measure will be regional standardized uptake value ratio (SUVR) values for 18F-MK-6240 using cerebellum as reference region. Kinetic modeling using Logan DVR method may also be employed. Multiple brain regions will be measured, with particular attention to medial temporal cortex structures such as hippocampus and entorhinal cortex

CONTACTS AND LOCATIONS:
Overall Officials: Jose A. Luchsinger, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share data with the data sharing platform of the NIA consortium named "Molecular Mechanisms of the Vascular Etiology of Alzheimer's disease (M2OVE-AD)" for data collection supported by grant RF1AG051556. This data sharing platform is called Synapse, and is managed by SAGE bionetworks. The main data from this protocol to be shared are summary values of brain Tau SUVR, demographics, and clinical variables such as diabetes status.
Supporting Information: Study Protocol
Time Frame: Data will be released twice a year to SAGE bionetworks for sharing.
Access Criteria: Synapse operates under comprehensive governance policies. These policies delineate Synapse users' rights and responsibilities. They also specify the rights and responsibilities of Sage Bionetworks and of the Synapse Access and Compliance Team (ACT).
URL: https://help.synapse.org/docs/

REFERENCES:
- [Background] Palta P, Rippon B, Tahmi M, Pardo M, Johnson A, Tomljanovic Z, He H, Laing KK, Razlighi QR, Teresi JA, Moreno H, Brickman AM, Kreisl WC, Luchsinger JA. Sex differences in in vivo tau neuropathology in a multiethnic sample of late middle-aged adults. Neurobiol Aging. 2021 Jul;103:109-116. doi: 10.1016/j.neurobiolaging.2021.03.007. Epub 2021 Mar 23. PMID 33894641
- [Result] Kreisl WC, Lao PJ, Johnson A, Tomljanovic Z, Klein J, Polly K, Maas B, Laing KK, Chesebro AG, Igwe K, Razlighi QR, Honig LS, Yan X, Lee S, Mintz A, Luchsinger JA, Stern Y, Devanand DP, Brickman AM. Patterns of tau pathology identified with 18 F-MK-6240 PET imaging. Alzheimers Dement. 2022 Feb;18(2):272-282. doi: 10.1002/alz.12384. Epub 2021 May 31. PMID 34057284